CLINICAL TRIAL: NCT06502808
Title: The Effect of Hyperbaric Oxygen Therapy on Oxidative Stress and Inflammation in Patients With Diabetic Foot Ulcers
Brief Title: Hyperbaric Oxygen Therapy in Diabetic Foot
Acronym: HBOTDF
Status: Completed | Type: Observational
Sponsor: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Modesto Gómez López, Doctor in Research in Medicine (Molecular Biology), School of Medicine, National Polytechnic Institute. Polytechnic Institute., National Polytechnic Institute, Mexico
Other Study IDs: CEI-CICS-038
Record Dates: First submitted 2024-06-20; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot Ulcer Neuropathic
Keywords: Gene expression; Hyperbaric oxygen therapy; Diabetic foot
MeSH Terms: conditions — Diabetic Foot | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — Series of 30 HBOT sessions of 60 minutes at 2 ATA in the hyperbaric chamber for five consecutive days per week.

SUMMARY:
This study seeks to assess changes in genes that are related to inflammation and oxidative stress in patients with type 2 Diabetes with diabetic foot treated with hyperbaric chamber

DETAILED DESCRIPTION:
Aims: Patients with an uncontrolled glycemic index develop a wide variety of pathologies associated with diabetes, such as diabetic foot ulcers (DFUs). Hyperbaric oxygen therapy (HBOT) is an adjunctive therapy used to help wound healing and prevent lower extremity amputations in this population. The aim of this study was to analyze the effect of HBOT on the gene expression of Super Oxide Dismutase 1 (SOD1), Super Oxide Dismutase 2 (SOD2), Glutathione Peroxidase (GPX2), and pro-inflammatory cytokines (TNFα, IL-1β, IL-12, IL-4, NLRP3) in patients with Wagner stage II-IV DFUs.

Methods: The effect of HBOT was evaluated in 15 patients that underwent 12 and 30 sessions in the hyperbaric chamber. Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR). In the analysis, qualitative variables are presented in frequencies and percentages, compared with the Chi-square test; quantitative variables according to the Shapiro-Wilk normality test, normally distributed variables are presented in means and standard deviation, compared with Student;s t-test, those related with ANOVA test; quantitative variables of free distribution are presented in medians and interquartile ranges, compared with Mann Whitney U-test, those related with Kruskall-Wallis test. Data analysis was carried out with SPSS version 23, Graph Pad Prisma. A value p < 0.05 was taken as statistical significance, 95%.

ELIGIBILITY:
Inclusion Criteria:

Men and women with diabetic foot and hyperbaric treatment. Ages 30-60 years. Signed informed consent form.

Exclusion Criteria:

* Patients with diabetic foot without presence of dermatologic lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men older than 18 years, with Diabetes type 2, residents of the CDMX, with diabetic foot with hyperbaric treatment, attended at the hospital of specialties in diabetes, secretary of health, accepted and signed the informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Gene expression of superoxide dismutase 1/ SOD1 | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  . Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Gene expression of superoxide dismutase 2 | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Glutathione Peroxidase (GPX2) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Interleukin-1β (IL-1β) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Interleukin-4 (IL-4) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Interleukin-12 (IL-12) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
NLRP3 inflammasome (NOD-, LRR- and pyrin domain-containing protein 3) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).
Tumor necrosis factor alpha (TNF-α) | The effect of the hyperbaric chamber was evaluated after sessions 12 and 30, each session lasting 60 minutes for five consecutive days per week, for a total of 6 weeks.
  Blood samples were collected and relative gene expression was assessed by quantitative real time polymerase chain reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Modesto Gómez López, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Godman CA, Chheda KP, Hightower LE, Perdrizet G, Shin DG, Giardina C. Hyperbaric oxygen induces a cytoprotective and angiogenic response in human microvascular endothelial cells. Cell Stress Chaperones. 2010 Jul;15(4):431-42. doi: 10.1007/s12192-009-0159-0. Epub 2009 Dec 1. PMID 19949909
- [Result] van Neck JW, Tuk B, Fijneman EMG, Redeker JJ, Talahatu EM, Tong M. Hyperbaric oxygen therapy for wound healing in diabetic rats: Varying efficacy after a clinically-based protocol. PLoS One. 2017 May 17;12(5):e0177766. doi: 10.1371/journal.pone.0177766. eCollection 2017. PMID 28545109
- [Result] undefined
- [Result] Dadmanesh M, Ranjbar MM, Ghorban K. Inflammasomes and their roles in the pathogenesis of viral hepatitis and their related complications: An updated systematic review. Immunol Lett. 2019 Apr;208:11-18. doi: 10.1016/j.imlet.2019.03.001. Epub 2019 Mar 1. PMID 30831142
- [Result] Hsieh CP, Chiou YL, Lin CY. Hyperbaric oxygen-stimulated proliferation and growth of osteoblasts may be mediated through the FGF-2/MEK/ERK 1/2/NF-kappaB and PKC/JNK pathways. Connect Tissue Res. 2010 Dec;51(6):497-509. doi: 10.3109/03008201003746679. Epub 2010 May 24. PMID 20497028
- [Result] Clokie M, Greenway AL, Harding K, Jones NJ, Vedhara K, Game F, Dhatariya KK. New horizons in the understanding of the causes and management of diabetic foot disease: report from the 2017 Diabetes UK Annual Professional Conference Symposium. Diabet Med. 2017 Mar;34(3):305-315. doi: 10.1111/dme.13313. Epub 2017 Jan 23. PMID 28029181
- [Result] Matchett GA, Martin RD, Zhang JH. Hyperbaric oxygen therapy and cerebral ischemia: neuroprotective mechanisms. Neurol Res. 2009 Mar;31(2):114-21. doi: 10.1179/174313209X389857. PMID 19298750
- [Result] Michalski D, Hartig W, Schneider D, Hobohm C. Use of normobaric and hyperbaric oxygen in acute focal cerebral ischemia - a preclinical and clinical review. Acta Neurol Scand. 2011 Feb;123(2):85-97. doi: 10.1111/j.1600-0404.2010.01363.x. PMID 20456243
- [Result] Calvert JW, Cahill J, Zhang JH. Hyperbaric oxygen and cerebral physiology. Neurol Res. 2007 Mar;29(2):132-41. doi: 10.1179/016164107X174156. PMID 17439697

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06502808/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06502808/ICF_001.pdf